CLINICAL TRIAL: NCT03401034
Title: The Influence of Lifestyle and Genetic Risk Factors, Circulating Inflammatory Biomarkers and Menopausal Hormone Therapy on Long-term Prognosis After Postmenopausal Breast Cancer
Brief Title: Influence of Lifestyle, Inflammatory Biomarkers, and Genetic Factors on Long-term Breast Cancer Prognosis
Status: Completed | Type: Observational
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: GermanCRC_ID76
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer; Breast Cancer Mortality; Breast Cancer Survival; Postmenopausal Breast Cancer; Lifestyle; Genetic Factors; Inflammation; Inflammatory Biomarkers; Hormone Therapy; Phytoestrogens
MeSH Terms: conditions — Breast Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nonfasting serum or plasma samples provided at recruitment and follow-up by the patients are stored at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MARIEplus study is a prospective cohort of breast cancer patients recruited into the MARIE (Mamma Carcinoma Risk factor InvEstigation) study, a population-based case-control study of breast cancer conducted in two German study regions, Hansestadt Hamburg and Rhine-Neckar-Karlsruhe (RNK) region. Participants were identified through participating clinics and the Hamburg cancer registry between January 1st, 2001 and September 30th, 2005 in Hamburg and between August 1st, 2002 and July 31st, 2005 in the RNK study region. Patients were aged 50-74 years at histologically confirmed primary invasive (stages I to IV) or in situ breast tumor (stage 0). Comprehensive information on demographic, socio-economic, and lifestyle factors was collected at multiple time points: at recruitment by a standardized face-to-face interview and at follow-up median 6 years as well as 11 years later using computer assisted telephone interview.

Vital status was assessed in 2009 and again in 2015 via the population registries and causes of death were obtained from death certificates and coded according to the 10th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-10).

Information on the clinical course was abstracted from medical records to verify clinical events either self-reported in follow-up interviews or reported by treating physicians.

The studies were approved by the ethics committee of the University of Heidelberg and the University of Hamburg and conducted in agreement with the Helsinki Declaration. Written informed consent was provided by all participants at baseline and during follow-up.

The primary objectives of this study are

* To assess the association of modifiable lifestyle factors and personal factors, including BMI, diet, physical activity, tobacco and alcohol use, menopausal hormone therapy, socioeconomic status, with breast cancer survival, overall and according to tumor type, after accounting for established prognostic factors.
* To examine the influence of genetic variants on breast cancer relapse and survival
* To assess the association of lifestyle factors and their changes in the course of survivorship on subsequent breast cancer prognosis.
* To assess the individual and combined association of inflammation/metabolic biomarkers as well as changes in their serum levels with subsequent breast cancer prognosis overall and according to tumor type.
* To assess whether and to what extent the associations between breast cancer prognosis and lifestyle factors and/or their changes are mediated by circulating biomarker levels.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Primary invasive (ICD-10 C50) (stage I-IV) or in-situ (ICD-10 D05) breast cancer
* 50 to 74 years at diagnosis
* Patients in the city and state of Hamburg in northern Germany and the Rhine-Neckar-Karlsruhe region in southern Germany
* German-speaking
* Physically and mentally ability to participate in a personal interview of about 90 minutes

Exclusion Criteria:

* Previous diagnosis of breast cancer

Ages: 50 Years to 74 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed primary invasive or in situ breast tumors aged 50-74 years at diagnosis recruited in the city and state of Hamburg or the Rhine-Neckar-Karlsruhe region
Sampling Method: Probability Sample
Enrollment: 3813 (Actual)
Dates: Start 2002-08-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality after breast cancer diagnosis | Median follow-up time 6 and 11 years
  Risk of mortality (all-cause, breast cancer specific)

SECONDARY OUTCOMES:
Risk of recurrence | Median follow-up time 6 and 11 years
  Risk of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Chang-Claude, Prof. Dr., Principal Investigator — German Cancer Research Center